CLINICAL TRIAL: NCT04437303
Title: Periprocedural Continuation Versus Interruption of Oral Anticoagulant Drugs During Transcatheter Aortic Valve Implantation (POPular PAUSE TAVI)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St. Antonius Hospital (Other)
Responsible Party: Principal Investigator, Jurriën M. ten Berg, MD, PhD, Professor dr., St. Antonius Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NL73805.100.20
Record Dates: First submitted 2020-05-19; First posted 2020-06-18 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Aortic Valve Disease; Aortic Valve Stenosis; Stroke; Bleeding; Vascular Complications; Myocardial Infarction; Thrombosis Embolism
Keywords: Transcatheter Aortic Valve Implantation (TAVI); Transcatheter Aortic Valve Replacement (TAVR); Aortic Valve Disease; Aortic Valve Stenosis; Stroke; Bleeding; Vascular Complications; Myocardial Infarction; Thrombosis Embolism; Heart Diseases; Oral Anticoagulation; Warfarin; Vitamin K Antagonist; Direct Acting Oral Anticoagulants; Protamine
MeSH Terms: conditions — Aortic Valve Disease; Aortic Valve Stenosis; Stroke; Hemorrhage; Myocardial Infarction; Embolism and Thrombosis; Heart Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuation of oral anticoagulants (Active Comparator)
  Interventions: Drug: Continuation of oral anticoagulants
- Interruption of oral anticoagulants (Active Comparator)
  Interventions: Drug: Interruption of oral anticoagulants

INTERVENTIONS:
Drug: Continuation of oral anticoagulants — Oral anticoagulant treatment will not be interrupted before the procedure.
  Arms: Continuation of oral anticoagulants
Drug: Interruption of oral anticoagulants — Peri-operative interruption of oral anticoagulants will be according to the Dutch guideline on antithrombotic therapy.
  * For direct oral anticoagulant users this will be in general 48 hours before the procedure, except for Dabigatran users with renal insufficiency: with estimated glomerular filtration rate 50-80 mL/min/1.73m^2 72 hours and with estimated glomerular filtration rate 30-50 mL/min/1.73m^2 96 hours before procedure.
  * For vitamin K antagonist users this will be 5 days for phenprocoumon and 3 days for acenocoumarol.
  * After the procedure oral anticoagulants will be resumed after 24 hours, if deemed safe by the treating physician.
  Arms: Interruption of oral anticoagulants

SUMMARY:
Transcatheter aortic valve implantation (TAVI) is a rapidly growing treatment option for patients with aortic valve stenosis. Stroke is a feared complication of TAVI, with an incidence of around 4-5% in the first 30 days. Up to 50% of patients undergoing TAVI have an indication for oral anticoagulants (OAC) mostly for atrial fibrillation. OAC use during TAVI could increase bleeding complications, but interruption during TAVI may increase the risk for thromboembolic events (i.e. stroke, systemic embolism, myocardial infarction). Recent observational data suggest that periprocedural continuation of OAC is safe and might decrease the risk of stroke. Beside the potential reduction of thromboembolic events, continuation of OAC is associated with an evident clinical ancillary benefit for patients and staff. Since periprocedural OAC interruption not infrequently leads to misunderstanding and potentially dangerous situations, when patients are not properly informed before hospital admission or may experience difficulties with the interruption regimen.

Hypothesis:

Periprocedural continuation of oral anticoagulants is safe and might decrease thromboembolic complications without an increase in bleeding complications at 30 days

ELIGIBILITY:
Inclusion Criteria:

* Planned transfemoral or transsubclavian transcatheter aortic valve implantation procedure
* Uses oral anticoagulation at screening
* Provided written informed consent

Exclusion Criteria:

Patients at high risk for thromboembolism for whom interruption of oral anticoagulants is no option, i.e.:

* Mechanical heart valve prosthesis
* Intracardiac thrombus
* < 3 months after venous thromboembolism
* < 6 months after transient ischemic attack or stroke in patients with atrial fibrillation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 858 (Actual)
Dates: Start 2020-11-25 (Actual); Primary Completion 2024-03-21 (Actual); Study Completion 2024-05-22 (Actual)

PRIMARY OUTCOMES:
Net adverse clinical events | 30 days
  A composite of cardiovascular mortality, all stroke, myocardial infarction, major vascular complications and type 2-4 bleeding complications at 30 days post TAVI as defined by the VARC-3 criteria

SECONDARY OUTCOMES:
Procedure related primary endpoints | 30 days
  Cardiovascular mortality, all stroke, myocardial infarction, major vascular complications and type 2-4 bleeding complications as defined by the VARC-3 criteria considered procedure related as adjudicated by the clinical event committee
Procedure related bleeding complications | 30 days
  Type 1-4 bleeding as defined by the VARC-3 criteria considered procedure related as adjudicated by the clinical event committee
Procedure related thromboembolic complications | 30 days
  All stroke (except haemorrhagic), TIA, myocardial infarction, systemic embolism (vascular complications: distal embolization (non-cerebral) from a vascular source) as defined by the VARC-3 criteria considered procedure related as adjudicated by the clinical event committee
Thromboembolic complications | 30 days
  All stroke (except haemorrhagic), TIA, myocardial infarction and systemic embolism (vascular complications: distal embolization (non-cerebral) from a vascular source) as defined by the VARC-3 criteria
Neurologic events | 30 days
  Overt CNS injury, covert CNS injury, neurologic dysfunction (acutely symptomatic) without CNS injury as defined by the VARC-3 criteria
Cerebrovascular events | 30 days
  All stroke and TIA as defined by the VARC-3 criteria.
Stroke | 30 days
  All stroke as defined by the VARC-3 criteria
Bleeding complications | 30 days
  Type 1-4 bleeding as defined by the VARC-3 criteria
Early safety | 30 days
  Freedom from all-cause mortality, all stroke, VARC type 2-4 bleeding, major vascular, access-related, or cardiac structural complication, acute kidney injury stage 3 or 4, moderate or severe aortic regurgitation, new permanent pacemaker due to procedure related conduction abnormalities, surgery or intervention related to the device as defined by the VARC-3 criteria
Clinical efficacy | 30 days
  Freedom from: all-cause mortality, all stroke, hospitalization for procedure- or valve-related causes, KCCQ Overall Summary Score <45 or decline from baseline of >10 point as defined by the VARC-3 criteria
All-cause death | 30 days
Cardiovascular death | 30 days
Quality of Life | 30 days and 90 days
  Assessed by Short Form(SF)-12, Kansas City Cardiomyopathy Questionnaire (KCCQ), and Toronto aortic stenosis quality of life questionnaire (TASQ)

OTHER OUTCOMES:
New York Heart Association class for heart failure | 30 days
Rehospitalisation | 30 days
Permanent pacemaker implantation | 30 days
Bleeding | 30 days
  As classified by Bleeding Academic Research Consortium (BARC) criteria

CONTACTS AND LOCATIONS:
Overall Officials: Jurriën M ten Berg, MD PhD, Principal Investigator — St. Antonius Hospital
Locations (22):
- Belgium (7):
  - A.S.Z. Hospital, Aalst
  - O.L.V. Hospital, Aalst
  - ZNA Middelheim, Antwerp
  - AZ Sint-Jan, Bruges
  - East Limburg Hospital, Genk
  - University Hospital Leuven, Leuven
  - AZ Delta, Roeselare
- Rigshospitalet Copenhagen, Copenhagen, Denmark
- University Hospital Galway, Galway, Ireland
- Azienda Sanitaria Universitaria Integrata di Trieste, Trieste, Italy
- National Institute of Cardiac Surgery and Interventional Cardiology, Luxembourg, Luxembourg
- Netherlands (11):
  - St. Antonius Ziekenhuis, Nieuwegein, Utrecht
  - Amsterdam UMC, Amsterdam
  - Amphia Hospital, Breda
  - UMC Groningen, Groningen
  - Leiden University Medical Center, Leiden
  - Maastricht UMC+, Maastricht
  - Radboud UMC, Nijmegen
  - Erasmus MC, Rotterdam
  - Haga Hospital, The Hague
  - UMC Utrecht, Utrecht
  - Isala, Zwolle

REFERENCES:
- [Derived] van Bergeijk KH, Overduin DC, Venema CS, van Ginkel DJ, van der Werf HW, van den Heuvel AFM, Voors AA, Wykrzykowska JJ, Ten Berg JM. Sex Differences in Transcatheter Aortic Valve Implantation Outcomes in Patients on Oral Anticoagulants: A Popular PAUSE TAVI SubAnalysis. J Am Heart Assoc. 2025 Nov 4;14(21):e043448. doi: 10.1161/JAHA.125.043448. Epub 2025 Oct 23. PMID 41128170
- [Derived] van Ginkel DJ, Bor WL, Aarts HM, Dubois C, De Backer O, Rooijakkers MJP, Rosseel L, Veenstra L, van der Kley F, van Bergeijk KH, Van Mieghem NM, Agostoni P, Voskuil M, Schotborgh CE, IJsselmuiden AJJ, Van Der Heyden JAS, Hermanides RS, Barbato E, Mylotte D, Fabris E, Frambach P, Dujardin K, Ferdinande B, Peper J, Rensing BJWM, Timmers L, Swaans MJ, Brouwer J, Nijenhuis VJ, Overduin DC, Adriaenssens T, Kobari Y, Vriesendorp PA, Montero-Cabezas JM, El Jattari H, Halim J, Van den Branden BJL, Leonora R, Vanderheyden M, Lauterbach M, Wykrzykowska JJ, van 't Hof AWJ, van Royen N, Tijssen JGP, Delewi R, Ten Berg JM; POPular PAUSE TAVI Investigators.; POPular PAUSE TAVI Investigators. Continuation versus Interruption of Oral Anticoagulation during TAVI. N Engl J Med. 2025 Jan 30;392(5):438-449. doi: 10.1056/NEJMoa2407794. Epub 2024 Aug 31. PMID 39216096